CLINICAL TRIAL: NCT06878040
Title: Effect of Baseline Ferritin Level on Iron Status in Male Elite Youth Rowers
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: WIOSŁA2023
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Inflammation; Iron Deficiency Anemias; Red Blood Cell
MeSH Terms: conditions — Inflammation; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Eppendorf tubes with serum.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The data of 16 trained men from the Polish Youth National Rowing. All athletes presented as medically fit, with no underlying health problems. In this cohort, baseline serum ferritin levels were considered, and the athletes were divided into two groups:

1. Serum ferritin <75 ng/ml (SF<75): n=9
2. Serum ferritin >75 ng/ml (SF>75): n=7

The rowing test was performed at the beginning of the preparatory phase of the annual training cycle (April), which is characterized by high volume and training load. After a 5-min of individual warm-up, the athletes performed a 2000-m exercise test on a rowing ergometer (Concept II, USA). Blood samples took from the cubital vein at three time points: before stress test (pre-exercise), one minute after the end of the test (post-exercise), and after a 1-hour recovery period (1h recovery).

Measurements ferritin, transferrin, hepcidin and interleukin-6 (IL-6) levels were determined using ELISA kits (SunRed Biotechnology Company). The iron levels were determined on the SPECTROstar Nano reader.

DETAILED DESCRIPTION:
The data of 16 trained men from the Polish Youth National Rowing. All athletes presented as medically fit, with no underlying health problems. In this cohort, baseline serum ferritin levels were considered, and the athletes were divided into two groups:

1. Serum ferritin <75 ng/ml (SF<75): n=9
2. Serum ferritin >75 ng/ml (SF>75): n=7

The rowing test was performed at the beginning of the preparatory phase of the annual training cycle (April), which is characterized by high volume and training load. After a 5-min of individual warm-up, the athletes performed a 2000-m exercise test on a rowing ergometer (Concept II, USA). Blood samples took from the cubital vein at three time points: before stress test (pre-exercise), one minute after the end of the test (post-exercise), and after a 1-hour recovery period (1h recovery).

Measurement: All determined parameters will be measured with the available equipment in the ZWKF laboratory in Gorzów Wielkopolski and using commercial assay kits. Measurements will be performed by the project contractors.

1. Polyethylene tubes (2.7ml) containing dipotassium ethylenediaminetetraacetic acid (EDTAK2) anticoagulant will be used for the following tests:

   (a) complete blood count (7 parameters) determined on the MYTHIC 18 hematology analyzer (Orphee Medical, Geneva, Switzerland). Red blood cell indices: RBC (Red Blood Cells), HGB (Hemoglobin), HCT (Hematocrit), MCV (Mean Corpuscular Volume), MCH (Mean Corpuscular Hemoglobin), MCHC (Mean Corpuscular Hemoglobin Concentration), RDW (Red Blood cells Distribution Width).
2. Polyethylene clotting activator tubes (9 ml) will be centrifuged to separate the morphotic elements from the serum using a centrifuge (3000 rpm for 10 min). The serum will be pipetted into several Eppendorf tubes, which will then be frozen (temp. -80 °C). All the following biochemical parameters will be determined from the extracted serum:

   1. using the ELISA method by the test manufacturer's instructions. The designations include the flowing parameters:

      * iron status parameters: hepcidin, transferrin , ferritin,
      * indicators of inflammation: IL-6.
   2. The iron levels be determined using the colorimetric method on the SPECTROstar Nano reader.
3. The lactate (La) concentration will be determined from the capillary blood immediately after collection using a commercially available kit (Dr. Lange, Germany).

Youth National Rowing Team of Poland The athletes' diets were completely analyzed before each exercise test by a nutritionist. Participants, with the help of a dietician who was available during meals on test days, filled out food diaries. The amount of energy, protein, carbohydrates, fats and fiber were then analyzed using a commercially available program.

The experiment was conducted in accordance with the Declaration of Helsinki. The study protocol was approved by the Ethical Committee of the Medical University of Poznan (decision no. 685/23 in 2023).

ELIGIBILITY:
Inclusion Criteria:

* Training experience a minimum of five years
* Minimum training time per week 240 minute
* Membership in the Youth National Rowing Team of Poland
* Completion of the 2000m ergometer test on two test dates

Exclusion Criteria:

* Taking other supplements containing anthocyanin compounds during the study period or a month earlier
* Antibiotic therapy
* Health problems

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Youth National Rowing Team of Poland
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Ferritin | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of ferritin [ng/mL]. ELISA method by the test manufacturer's instructions
Iron | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  The iron level [µg/dL] will be determined using the colorimetric method on the SPECTROstar Nano reader.
Interleukin-6 (Il-6) | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of IL-6 [ng/L]. ELISA method by the test manufacturer's instructions
Hepcidin | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of hepcidin [ng/mL]. ELISA method by the test manufacturer's instructions
Transferrin | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of transferrin [mg/mL]. ELISA method by the test manufacturer's instructions
The Blood morphology - RBC (Red Blood Cells) | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  RBC (Red Blood Cells) [106 × µL-1] determined on the MYTHIC 18 hematology analyzer (Orphee Medical, Geneva, Switzerland).
The Blood morphology- HGB (Hemoglobin) | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  HGB (Hemoglobin) [g/dL] determined on the MYTHIC 18 hematology analyzer (Orphee Medical, Geneva, Switzerland).
The Blood morphology- HCT (Hematocrit) | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  HCT (Hematocrit) [%]determined on the MYTHIC 18 hematology analyzer (Orphee Medical, Geneva, Switzerland).
The Blood morphology- MCV (Mean Corpuscular Volume) | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  MCV (Mean Corpuscular Volume)[fl] determined on the MYTHIC 18 hematology analyzer (Orphee Medical, Geneva, Switzerland).
The Blood morphology- MCH (Mean Corpuscular Hemoglobin) | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  MCH (Mean Corpuscular Hemoglobin) [pg] determined on the MYTHIC 18 hematology analyzer (Orphee Medical, Geneva, Switzerland).
The Blood morphology- MCHC (Mean Corpuscular Hemoglobin Concentration) | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  MCHC (Mean Corpuscular Hemoglobin Concentration) [g x dL-1] determined on the MYTHIC 18 hematology analyzer (Orphee Medical, Geneva, Switzerland).
The Blood morphology- RDW (Red Blood cells Distribution Width) | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  RDW (Red Blood cells Distribution Width) [%] determined on the MYTHIC 18 hematology analyzer (Orphee Medical, Geneva, Switzerland).

SECONDARY OUTCOMES:
Antropometric characteristic - height | Day 1 after overall fast
  Prior to the exercise test, the investigators measured the anthropometric parameters, including height (Seca 213 Hamburg, Deutschland) [cm]
Antropometric characteristic - weight | Day 1 after overall fast
  Prior to the exercise test, the investigators measured the anthropometric parameters, including weight (Tanita BC 418 MA, Tanita Corporation, Tokyo, Japan) [kg]
Food record - energy | Day before the Day 1, in the morning at Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: energy [kcal]
Food record - protein | Day before the Day 1, in the morning at Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: protein [g]
Food record - carobhydrates | Day before the Day 1, in the morning at Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: carbohydrates [g]
Food record - fiber | Day before the Day 1, in the morning at Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: fiber [g]
Food record - fat | Day before the Day 1, in the morning at Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: fat [g]

CONTACTS AND LOCATIONS:
Locations (1):
- Poznań University of Physical Education,, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No